CLINICAL TRIAL: NCT07172373
Title: Safety and Efficacy of Antegrade Flexible Ureteroscopy-Assisted Percutaneous Nephrolithotomy for Staghorn Calculi: A Prospective Multicenter Clinical Study
Brief Title: Safety and Effectiveness of Antegrade Flexible Ureteroscopy-Assisted Percutaneous Nephrolithotomy for Staghorn Calculi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Tianjin Medical University General Hospital (Other); Peking University People's Hospital (Other); First Hospital of China Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Tsinghua Changgeng Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The Affiliated Hospital of Qingdao University (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 062/2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Urolithiasis; Renal Stones
Keywords: Percutaneous nephrolithotomy; Antegrade flexible ureteroscopy; Staghorn calculi; Stone branch number
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Staghorn Calculi

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Because of the inherent differences between the two interventions, blinding of patients and surgeons is not feasible. Postoperative imaging (CT) will be evaluated by radiologists blinded to treatment allocation, and clinical outcomes will be assessed by investigators who were not involved in the surgeries and remained unaware of the intervention. In addition, statistical analyses will be conducted in a blinded manner, with analysts kept unaware of group assignments until all analyses and interpretations are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antegrade flexible ureteroscopy-assisted PCNL (Experimental): antegrade flexible ureteroscopy-assisted PCNL
  Interventions: Procedure: antegrade flexible ureteroscopy-assisted PCNL
- single PCNL (Other): single PCNL
  Interventions: Procedure: single PCNL

INTERVENTIONS:
Procedure: antegrade flexible ureteroscopy-assisted PCNL — antegrade flexible ureteroscopy-assisted PCNL
  Arms: antegrade flexible ureteroscopy-assisted PCNL
Procedure: single PCNL — single PCNL
  Arms: single PCNL

SUMMARY:
Objective This study aims to evaluate the safety and efficacy of antegrade flexible ureteroscopy-assisted PCNL for the treatment of staghorn calculi, compared with standard PCNL.

Methods This prospective, multicenter, randomized controlled trial plans to enroll 420 patients with staghorn calculi, randomly assigned into two groups: the experimental group (antegrade flexible ureteroscopy-assisted PCNL, n=210) and the control group (standard PCNL, n=210). The primary endpoint is stone-free rate (defined as no residual fragment ≥2 mm on postoperative CT). Secondary endpoints include operative time, number of percutaneous tracts, rate of secondary procedures, hemoglobin decrease, postoperative complications (Clavien-Dindo classification), and length of hospital stay. All patients will undergo CT evaluation on postoperative day 2. Subgroup analysis will be performed according to the number of stone branches (≥5 vs <5).

DETAILED DESCRIPTION:
Background Renal calculi are among the most common diseases in urology. Current treatment options include extracorporeal shock wave lithotripsy (ESWL), flexible ureteroscopic lithotripsy, and percutaneous nephrolithotomy (PCNL). For renal stones ≥2 cm, PCNL is the recommended first-line treatment.

However, because of the large stone burden and the involvement of multiple calyces, it is often difficult to achieve complete clearance with a single PCNL session. Excessive angulation of the nephroscope may increase the risk of infundibular tears and bleeding, and stones located in parallel or narrow infundibula may be difficult to access, reducing the one-stage stone-free rate. To improve outcomes, several strategies have been adopted:

Multiple percutaneous tracts: Establishing additional tracts allows access to calyces unreachable from the primary tract and increases stone-free rates. However, this also increases the risks of bleeding, infection, and injury to the kidney or adjacent organs. In addition, expansion of the first tract may cause perirenal hematoma or morphological changes due to urine extravasation, making subsequent punctures more challenging. Multiple tracts also prolong postoperative recovery and increase hospitalization costs. Staged procedures: The first PCNL session removes stones in the renal pelvis and accessible calyces, while residual stones are addressed in a second-stage retrograde ureteroscopy. This reduces the risks compared with multiple tracts, but prolongs the treatment cycle and increases costs. Endoscopic combined intrarenal surgery (ECIRS) with modified patient positions: Positions such as the modified supine split-leg, lateral decubitus, or female-specific "Galdakao-modified supine Valdivia" allow simultaneous use of ureteroscopic and percutaneous approaches. This combines the efficiency of PCNL with the wide access angle of ureteroscopy, reduces the need for repositioning under anesthesia, and facilitates intraoperative monitoring. However, it requires two surgical teams, duplicate equipment, and high coordination, which may prolong operative time.

Previous studies suggest that combining single-tract PCNL with flexible ureteroscopy and holmium laser lithotripsy may be an ideal approach for staghorn stones. While antegrade cystoscopic lithotripsy accommodates thicker fibers and offers faster irrigation and clearer visualization, the larger diameter of the cystoscope limits its passage through the ureter, risking residual fragments. Recently, antegrade flexible ureteroscopy-assisted PCNL has been attempted, but most studies are small retrospective series or case reports. The limited adoption may be due to the high purchase and repair costs of reusable flexible ureteroscopes. The development of single-use ureteroscopes has largely overcome these barriers, providing a foundation for multicenter prospective studies.

Based on this background, a multicenter clinical study of antegrade flexible ureteroscopy-assisted PCNL for staghorn calculi has important clinical value. Our preliminary work showed that when the number of stone branches was ≥5, the need for multiple tracts and staged procedures increased, while operative time was prolonged, hospital stay was longer, and the stone-free rate was reduced. We therefore further compared the efficacy of standard PCNL and antegrade flexible ureteroscopy-assisted PCNL stratified by stone branch number.

Objective To evaluate the safety and efficacy of antegrade flexible ureteroscopy-assisted PCNL in the treatment of staghorn calculi, compared with standard PCNL.

Study Overview Design This is a prospective, multicenter clinical study. Population

Inclusion criteria:

Diagnosis of staghorn calculi confirmed by non-contrast CT. Age ≥18 years. General condition suitable for surgery. Ability to understand and voluntarily sign informed consent.

Exclusion criteria:

Solitary kidney or congenital anomalies (e.g., horseshoe kidney, ectopic kidney). Severe preoperative pyelonephritis. Psychiatric illness or lack of cooperation. Uncontrolled comorbidities (e.g., diabetes, hypertension) contraindicating surgery. Coagulation disorders. Investigator's judgment of unsuitability.

Withdrawal criteria:

Subject withdrawal: refusal to continue or loss to follow-up. Investigator withdrawal: complications making continuation unsafe, or poor compliance.

Sample size and grouping

A total of 420 patients will be enrolled across 14 centers (30 per center). Patients will be randomized into two groups:

Experimental group: antegrade flexible ureteroscopy-assisted PCNL (n=210). Control group: standard PCNL (n=210).

Procedures All patients will undergo preoperative urine culture. Infected patients will receive targeted antibiotics until negative. Surgery will be performed under general anesthesia with tracheal intubation.

Standard PCNL group: Residual stones inaccessible through the primary tract will be managed by establishing a second or third tract.

Antegrade flexible ureteroscopy-assisted PCNL group: Residual stones will first be managed using a flexible ureteroscope introduced via the established tract. The Tianjin Institute of Urology (TJIU) technique will be adopted, systematically inspecting all calyces and the ureter. Additional tracts will be created only if necessary.

At the end of surgery, a double-J stent and nephrostomy tube will be placed. Postoperative evaluation： Stone-free rate (no residual fragments ≥2 mm on CT on postoperative day 2). Operative time (from tract establishment to nephrostomy placement). Complications (Clavien-Dindo classification). Secondary procedures. Postoperative fever. Length of hospital stay. Subgroup analysis will be conducted based on the number of stone branches (≥5 vs <5).

Endpoints Primary endpoint: Stone-free rate. Secondary endpoints: surgeon-perceived smoothness of operation, treatment satisfaction, rate of secondary procedures, operative time, number of tracts, hemoglobin decrease, length of hospital stay, postoperative complications.

Adverse Events

Definitions:

Adverse event (AE): any unfavorable medical occurrence after treatment, not necessarily causally related.

Serious adverse event (SAE): hospitalization, prolonged hospitalization, disability, life-threatening condition, death, or congenital anomaly.

Severity:

Mild: tolerable, no specific treatment needed. Moderate: requires intervention, directly affects recovery. Severe: life-threatening, fatal, or disabling, requiring emergency treatment.

Reporting:

All AEs/SAEs will be documented in case report forms with onset, presentation, management, and outcome. SAEs will be reported within 24 hours to the sponsor, ethics committee, and regulatory authorities.

Statistical Analysis This randomized, open-label, multicenter trial uses stone-free rate (CT on day 2, no fragments ≥2 mm) as the primary outcome. Based on preliminary data (stone-free rate ~52% for PCNL and ~71% for antegrade flexible ureteroscopy-assisted PCNL), sample size was calculated with 90% power and α=0.025, requiring 157 patients per group. Allowing for 20% attrition, 210 patients per group (420 total) will be enrolled.

Data will be analyzed using R software (version 4.1.2). Continuous variables will be expressed as mean ± SD, categorical variables as frequencies and percentages. Student's t-test, chi-square test, or Fisher's exact test will be used as appropriate. Two-sided p-values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Staghorn calculi confirmed by non-contrast CT of the urinary system; Age ≥18 years; General condition suitable for surgical treatment; Ability to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

Solitary kidney or congenital anomalies (such as horseshoe kidney or ectopic kidney); Patients with severe preoperative pyelonephritis; Patients with psychiatric disorders or unwilling to cooperate; Patients with uncontrolled diabetes or hypertension who cannot tolerate surgery; Patients with coagulation disorders; Patients deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Immediately stone-free rate (SFR) | On postoperative day 2, a non-contrast CT of the urinary system will be performed, and the absence of residual fragments larger than 2 mm will be defined as stone-free.
  defined as no residual fragment ≥2 mm on postoperative CT

SECONDARY OUTCOMES:
Operative time | From the establishment of the first percutaneous renal tract to the placement of the final nephrostomy tube.
  Operative time
Duration of hospital stay | Up to 3 months.
  Duration of hospital stay
Complications | Up to 3 months.
  Complications

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not share to other researchers as ethical issues.